CLINICAL TRIAL: NCT04043182
Title: ULTRASOUND FOR LOCAL FAT TREATMENT: A RANDOMIZED AND DOUBLE-BLIND CLINICAL TEST, CONTROLLED BY PLACEBO
Brief Title: EFFECTIVENESS OF ULTRASOUND FOR LOCAL FAT TREATMENT
Acronym: n
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: São Paulo State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SaoPSU_univar
Record Dates: First submitted 2019-07-12; First posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Fat Burn

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group control (No Intervention): You will not receive any type of intervention
- treatment group (ultrasound) (Experimental): Will perform protocols of 10 sessions of ultrasound in the region of abdomen
  Interventions: Procedure: ultrassound
- placebo group (Placebo Comparator): It will perform protocols of 10 sessions of ultrasound in the region of abdomen, but the apparatus will be with zero intensities
  Interventions: Procedure: ultrassound

INTERVENTIONS:
Procedure: ultrassound — The treatment protocol will consist of 10 sessions, lasting 20 minutes. The energy level corresponding to 59 J / cm2 (177 J / cm2) and frequency of 3 MHZ, applied in the anterior region of the abdomen, in a quadrant previously delimited with a ballpoint pen, will be used. The flanks (lateral of the abdomen) will not be treated.
  Arms: placebo group; treatment group (ultrasound)

SUMMARY:
It's evident that the literature shows good results on the use of aesthetic ultrasound in the treatment of localized fat, however, little has been explored so far, about possible psychological influences of this method and therefore, it is believed that it is pertinent to elaborate studies that include a placebo group, in order to measure the real effects from the exclusive application of ultrasound. Therefore, the objective of this study will be to verify the influence of the application of aesthetic ultrasound in the treatment of localized fat, using for both clinical, biochemical and functional parameters.

DETAILED DESCRIPTION:
There will be included 30 participants, female gender, communities between 18 and 30 years, apparently Saudi, local abdominal fat, located in three groups: control (n = 10), experimental (n = 10) and placebo (n = 10) . Or group control não recebeu nenhum type of intervention. No experimental group, 10 sessões de ultrassom (Skinner brand, São Paulo) will be carried out in the previous region for 20 minutes. No placebo group will be applied ultrassom (Skinner brand, São Paulo), pormem com zerada intensities. Anthropometric avaliação e of dobras cutâneas will be carried out at this time before applying the treatment protocol. As skin folds will be measured by means of adipometers.

ELIGIBILITY:
Inclusion Criteria:

* Additional inclusion criteria included body mass index (BMI) equal to or less than 25.0 kg / m2
* Adipose tissue thickness 2.6 cm or more in the treatment region;
* Preserved elasticity and local tissue integrity;
* In addition, participants had to agree not to change their daily routines during the study.

Exclusion Criteria:

* Pregnancy.
* Breastfeeding;
* History of liposuction;
* Lipolysis by injection therapy;
* Abdominoplasty or surgery in the treatment region;
* Weight reduction medication;
* Recent surgery in the last 12 months;
* Implantable electrical device;
* Neurosurgical deviation;
* Hernia;
* Sensory loss or dysesthesia in the treatment region;
* Cancer;
* Circulation problems;
* Or chronic systemic disease such as diabetes or metabolic syndrome.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-06-29 (Actual); Primary Completion 2019-09-25 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
change abdominal circumference (centimeters-cm), before and after intervention | before (day 0) and post protocol (post 8 weeks)
  To measure values corresponding to the waist / quadrile ratio, metric phyta will be used, which will collect measurements in centimeters (cm). Assim, at waist circumference, it will be measured at umbigo height.
change blood analysis (milligrams per decilitre-mg/dl ) before and after intervention | before (day 0) and post protocol (post 8 weeks)
  A biochemical analysis will be carried out with the use of soro from blood collection in the antecubital vein, collected at a quantity of 10 mL as participants in the jejum study did not start and end the treatment as ultrassom. As shown below, BIOPLUS 2000 semi-automatic biochemical method will be evaluated for a dosage of parameters such as Triglycerides, Total Cholesterol, High Density Lipoprotein - HDL and Baixa Densidade Lipoprotein Estimates - LDL and Baixíssima Densidade Lipoprotein - VLDL through calculation formula Friedewald As dosagens will be carried out not the Laboratory of Biochemistry of the University Center of Vale do Araguaia - UNIVAR).
weight (centimeters-cm) | before (day 0)
  stadiometer (Sanny, American Medical do Brasil, São Paulo, Brazil).

SECONDARY OUTCOMES:
anthropometric characteristics anthropometric characteristics, photometry and personal satisfaction | before (day 0)
  It will be measured by meio de uma meio de uma balança (Tanita BC554, Iron Man / Inner Scaner, Tanita, Illinois, United States) and a stadiometer (Sanny, American Medical do Brasil, São Paulo, Brazil). In this way, the height will be measured in centimeters and the weight in kilograms.
change photometry - reduction of waist measurements before and after intervention | before (day 0) and post protocol (post 8 weeks)
  A photograph will be taken with a professional camera of Canon Brand Powershot Sx530 Hs, with a fixed focal length and constant lighting.
personal satisfaction of the participants treated before and after intervention | before (day 0) and post protocol (post 8 weeks)
  A satisfação pessoal will be measured by means of a questionnaire, the objective of which will be to investigate these variables in a subjective way. Assim, the participants will be instructed to trace a 10 cm analog visual scale between two extremes, being 0 or "minimum possível" and 10 indicating "or more possível" for each classification. The satisfaction scale ranges from zero to ten.

CONTACTS AND LOCATIONS:
Locations (1):
- Jaqueline Lopes, Barra do Garças, Mount, Brazil

IPD SHARING:
Plan to Share IPD: No